CLINICAL TRIAL: NCT05164406
Title: Impact of Blood Salvage Therapy During Oncologic Liver Surgeries on Allogenic Transfusion Events, Survival and Recurrence
Brief Title: Impact of Blood Salvage Therapy on Outcomes After Oncologic Liver Surgery
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-2534
Record Dates: First submitted 2021-12-07; First posted 2021-12-20 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Liver Neoplasms
Keywords: Blood salvage therapy; Oncologic liver surgery
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With blood salvage: Patients undergoing oncologic liver surgery with systematic use of blood salvage therapy
  Interventions: Procedure: Blood salvage therapy
- Without blood salvage: Patients undergoing oncologic liver surgery without any blood salvage therapy

INTERVENTIONS:
Procedure: Blood salvage therapy — In the blood salvage group, blood is systematically given back when the minimal amount of blood loss required for reprocessing is met
  Groups: With blood salvage

SUMMARY:
A before and after trial comparing the systematic use of blood salvage therapy with leucocyte filter during oncologic liver resections. Recurrence, survival, allogenic transfusion rates and surgical outcomes are compared with a representative historic cohort.

DETAILED DESCRIPTION:
Blood salvage therapy in oncologic liver surgery is seldom used based on unproven concerns about the safety of the technique regarding potential cancer dissemination or recurrence. Nevertheless, the technique has proven advantages in other surgical settings regarding the allogenic transfusion outcomes. Allogenic blood transfusion has been scientifically proven to worsen prognosis in oncologic surgery. This study compares a cohort of patients systematically exposed the blood salvage therapy to one comparable cohort without the therapy and outcomes regarding transfusion rates, post-operative Hb measurement, recurrence, overall survival, and post-operative adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adult Oncologic liver surgery scheduled in our institution

Exclusion Criteria:

* Condition precluding consent for trial Pregnancy

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults undergoing liver surgery for any cancer in our institution between january 2018 and August 2019 (blood salvage group) and patients who underwent liver surgery without blood salvage between 2011 and 2018 (control group)
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Recurrence free survival | 18 months
Overall survival | 18 months
Transfusion | Up to 30 days after surgery
  Allogenic blood products requirements

CONTACTS AND LOCATIONS:
Overall Officials: Yves Collin, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lugassy L, Marion S, Balthazar F, Cheng Oviedo SG, Collin Y. Impact of blood salvage therapy during oncologic liver surgeries on allogenic transfusion events, survival, and recurrence: an ambidirectional cohort study. Int J Surg. 2024 Jun 1;110(6):3392-3400. doi: 10.1097/JS9.0000000000001458. PMID 38666789